CLINICAL TRIAL: NCT01380795
Title: Biological Study of Feasibility Concerning the Research for Mutation of the Gene of EGFR and for K-Ras in Circulating Tumoral Cells(CTCs) of the Patients Carriers of Metastatic Non Small Cells Bronchial Carcinomas
Brief Title: Feasibility of the Research for Mutation of K-ras and EGFR in CTCs From Metastatic Non Small Cells Bronchial Carcinomas
Acronym: CTC-Poumon
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0416-1cobr10
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2014-09

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: non-small cell lung cancer carcinoma; circulating tumor cells; EGFR; K-ras
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Circulating Tumor Cell (Other): blood sample CTC monitoring and CTC EGFR/K-ras status determination
  Interventions: Biological: CTC

INTERVENTIONS:
Biological: CTC — every two cures of a standard chemotherapy patients will be taken sample of blood to monitor CTC presence and EGFR/ K-ras status of that CTC

SUMMARY:
The knowledge concerning the biology of the human tumors do not stop widening, in particular concerning the molecular mechanisms at the origin of the process of carcinogenesis and its ability to become perpetual. The identification and the increasing knowledge of these abnormalities allowed during these last years the development of therapeutic strategies targeting specifically the molecular pathways involved in the carcinogenesis. It quickly lead to numerous therapeutic successes in association with conventional chemotherapy, allowing a better individualization of the treatment according to the biological characteristics of the tumor of the patient.

However such therapeutics are effective only if the patients carries specific genomic mutations making necessary the systematic research for one kind of mutation.

The problem is that currently the mutational status is frequently made on the tissue resulting from the initial tumor biopsy, and as it is not excluded that the evolution of the biology of the metastasis reports a different genomic status, the only theoretical solution is then to make biopsy systematically on metastasis, what is not always technically possible. The problem still complicates when the investigators know that the biology of the tumor may evolve in time, particularly under treatment, with appearance of chemotherapy resistant clones. The monitoring of the genomic status of the tumor thus appears to be a crucial stake in the next years in cancer research as far as the efficiency of numerous therapeutic targeted put at the disposal of the clinician, depends on it largely. The repeated access to tumor tissue, during the follow-up of the patient in treatment, seems from then on indispensable to guide prematurely the therapeutics, in particular by stopping a targeted therapeutics which the investigators know that it is not any more going to be effective, and so avoiding exposing the patient to useless toxicity of a treatment often extremely expensive, and of which usage should have to be reserved to patient who could respond to it.

The access to the circulating tumor cells in the blood of patients is a repeatable, not invasive technique (blood test) and henceforth accessible thanks to a technique using a magnetic sorting of the tumor cells selected by an antibody directed against the tumor antigen EpCAM. This new technology (CellSearch, Veridex system) totally standardized and automated, allows from a total sample of blood of the patient, to determine the quantity of circulating tumor cells (CTC).The number of CTC seems to constitute in recent studies, a powerful prognosis tool at the moment diagnosis, but also during treatment, according to its decrease or not under chemotherapy. In United States, the Food and Drug Administration (FDA) recently approved the use of this system for the quantification of the CTCs in the care of the patients affected by breast, colon, and prostate cancer. The CellSearch system will probably become in the future years an indispensable tool to help the clinicians to encircle better the prognosis of their patient. This technology already allows to realize besides a quantification, the isolation of viable CTCs, from which the genetic material can be extracted, amplified thus potentially analyzed. The investigators thus see all the interest which such a device can represent in the non invasive monitoring of the patients under treatment targeting molecular abnormality susceptible to evolve in time. The investigators thus propose to study thanks to the system CellSearch the feasibility of the research for the mutation of K-Ras and EGFR in the CTC of patients carriers of a metastatic non small cells bronchial carcinoma.

Secondly, the investigators research will be interested in the possible conflicts existing between the primitive tumor and the CTCs for the various popular mutations. In case of feasibility of the method, and the good initial concordance between the genomic status of the CTCs and that of the tumor, the investigators shall describe the genomic evolution under treatment monitoring the CTCs of the patients under targeted therapeutics. The investigators shall describe then if the premature observation of modification precedes the appearance of an effective resistance in treatments.

ELIGIBILITY:
Inclusion Criteria:

1. men and women
2. age over 18 y.o.
3. signed informed consent form.
4. Patients barriers of Non-small Cell Lung Cancer Metastatic
5. chemotherapy non yet begun
6. patients barrier of CTC
7. Research for mutation of EGFR and Kras made on the primitive tumor
8. Man and woman old enough to procreate under effective contraceptives

Exclusion Criteria:

1. small cells bronchial cancer
2. Non metastatic bronchial cancer
3. Absence of detectable CTC at the patient
4. Private individuals of freedom or under tutelage (including legal guardianship)
5. Incapacity to sign the inform consent form or psychiatric, behavioural disorders or geographical situation precluding the follow-up of the protocol
6. Pregnancy, lactating or refusal of the contraception for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03-09 (Actual); Primary Completion 2011-03-09 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
search for the mutation of EGFR and Kras in the CTC of the patient | september 2012 (anticpated) up to 2 years

SECONDARY OUTCOMES:
Compare EGFR/ K-ras status between CTC and the primitive tumor | september 2012 (anticipated) up to 2 years
Monitoring of the mutations of EGFR / K-ras in the CTC of the patients during treatment | september 2012 (anticipated) up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France